CLINICAL TRIAL: NCT00847158
Title: A Randomized, Double-Masked Clinical Trial of Phacoemulsification Compared With Phacoemulsification and Micro-Bypass Stent Implantation in Patients With POAG
Brief Title: A Clinical Trial of Phacoemulsification Versus Phacoemulsification & the iStent Implantation in POAG Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Responsible Party: Antonio Fea, University of Turin, Italy
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: iStent Washout study
Record Dates: First submitted 2009-02-18; First posted 2009-02-19 (Estimated); Last update posted 2009-02-19 (Estimated); Status verified 2009-02

CONDITIONS: Primary Open Angle Glaucoma and Cataracts
Keywords: POAG; Combination glaucoma & cataract procedure; trabecular micro-bypass stent; iStent
MeSH Terms: conditions — Glaucoma, Open-Angle; Cataract | interventions — Phacoemulsification; Cataract Extraction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): phacoemulsification alone
  Interventions: Procedure: phacoemulsification alone
- 2 (Active Comparator): phacoemulsification and implantation of the iStent® trabecular micro-bypass stent
  Interventions: Device: iStent Trabecular Micro-Bypass Stent

INTERVENTIONS:
Procedure: phacoemulsification alone — phacoemulsification alone
  Other Names: cataract surgery; Phaco
  Arms: 1
Device: iStent Trabecular Micro-Bypass Stent — phacoemulsification and implantation of the iStent® trabecular micro-bypass stent
  Other Names: iStent, Trabecular micro-bypass stent, GTS100L, GTS100R
  Arms: 2

SUMMARY:
This was a prospective, double-masked, 15-month clinical trial comparing efficacy of phacoemulsification alone to combined phacoemulsification and implantation of the iStent® trabecular micro-bypass stent in patients with primary open-angle glaucoma.

DETAILED DESCRIPTION:
This was a prospective, randomized open-label study of 36 patients with POAG scheduled to undergo phacoemulsification with intraocular lens implantation ("cataract surgery"). Patients were randomized 2:1 to receive either cataract surgery alone (control group) or cataract surgery and iStent implantation (combined surgery group).

Implantation of the study stent occurred after cataract extraction and IOL insertion using the same small, temporal, clear-corneal incision (approximately 3 mm) used to perform phacoemulsification and IOL placement. The study stent was guided into Schlemm's canal using ab-interno gonioscopy (using a Swan-Jacobs gonioscope). (Figure 1) If no complications occurred during phacoemulsification, acetylcholine was injected in the anterior chamber after the IOL implantation to constrict the pupil. The anterior chamber was then filled with a viscoelastic agent to reform the anterior chamber and provide more clearance in the angle.

The anterior chamber was traversed with the applicator (the implant was on the tip of applicator) and the trabecular meshwork located. The leading edge of the device was gently slid through the trabecular meshwork and into Schlemm's canal at the nasal position (3 to 4 o'clock for the right eye; 9 to 8 o'clock for the left eye) with the tip of the implant directed inferiorly. If difficulty was encountered with the insertion at the primary location, we tried inserting about 0.5 clock hour inferiorly; and continued to move inferiorly as needed for subsequent attempts. Next, the device was released by pushing the button on the applicator, position of the stent was verified and the applicator was withdrawn.

The patients were instructed to discontinue all glaucoma medications after surgery. Standard post cataract extraction antibiotic and anti-inflammatory drug regimen was prescribed. Target pressure for each patient was determined prior to study entry. Following the assigned procedure, any patient with an IOP (as measured between 8 and 10 AM) that was greater than 2 mm Hg over their target was instructed to return twice in the following three days for re-measurement of their IOP. If the patient's IOP was > 2 mm Hg over their target pressure, ocular hypotensive agents were added. The medications were added in a pre-set schedule, with beta-blockers first, angiotensin-converting enzyme (ACE) inhibitors second, and prostaglandins third. If, however, on the third consecutive visit the patient's IOP was within 2 mm Hg of target, patient re-entered the normal visit schedule. Investigators were masked to treatment assignment both when measuring IOP and when determining when or if to add medications.

ELIGIBILITY:
Inclusion Criteria:

* a previous diagnosis of POAG
* an IOP of > 18 mm Hg at three separate visits if on one medication, or subjects on at least two medications with uncontrolled IOP on three separate visits.
* all patients were deemed likely to follow surgeon instructions and were able to give informed consent.

Exclusion Criteria:

* any glaucoma diagnosis other than POAG
* the presence of peripheral anterior synechiae (PAS)
* a cloudy cornea likely to inhibit gonioscopic view of the angle
* any previous ocular surgery
* history of trauma or ocular surface disease
* the presence of peripheral anterior synechiae (PAS)
* a cloudy cornea likely to inhibit gonioscopic view of the angle

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2006-12; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Primary outcomes included IOP and reduction in medication use. | 15 month

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Fea, MD, Principal Investigator — University of Torino

REFERENCES:
- [Derived] Fea AM, Consolandi G, Zola M, Pignata G, Cannizzo P, Lavia C, Rolle T, Grignolo FM. Micro-Bypass Implantation for Primary Open-Angle Glaucoma Combined with Phacoemulsification: 4-Year Follow-Up. J Ophthalmol. 2015;2015:795357. doi: 10.1155/2015/795357. Epub 2015 Oct 26. PMID 26587282